CLINICAL TRIAL: NCT03765151
Title: The Effectiveness of Low-level Laser Therapy as an Adjunct Strategy in Orthodontic Retention for Periodontal-compromised Patients
Brief Title: The Effectiveness of Low-level Laser Therapy in Orthodontic Retention for Periodontal-compromised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HKUCTR-2390
Record Dates: First submitted 2018-11-21; First posted 2018-12-05 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Orthodontics; Periodontal Diseases
Keywords: low-level laser therapy; orthodontic retention; periodontal disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT group (Experimental): Low-level laser therapy and orthodontic retention
  Interventions: Device: low-level laser therapy; Other: orthodontic retention
- control group (Placebo Comparator): orthodontic retention and no laser treatment.
  Interventions: Other: orthodontic retention

INTERVENTIONS:
Device: low-level laser therapy — LLLT will be performed by a diode gallium-aluminum-arsenide (Ga-Al-As) laser with a 940-nm wavelength (Ezlase; Biolase Technology Inc., Irvine, CA) and delivered by a quadrant-sized probe which cover the region from the central incisor to the first molar on the test side. The laser probe will be 1 cm from the soft tissue around the test tooth at the gingival margin and alveolar mucosa covering the root area using a setting of 800 milliwatt in a continuous wave. Each tooth will receive 30 seconds of exposure, with no more than 8.6 J/cm2 of energy delivered. In addition, a spot-size laser probe will be applied for 30 seconds 5 mm from the cervical dentin with an output power of 700 milliwatt to reduce tooth sensitivity.
  Arms: LLLT group
Other: orthodontic retention — All participants included will wear fixed lingual retainer and removable retainers in the post-orthodontic retention period and their previous orthodontic treatment will be carried out by one operator using preadjusted appliances with bonded 0.022×0.028-inch2 brackets/buccal tubes and 0.014-inch Nickel Titanium (NiTi) archwires as the first archwires.

SUMMARY:
The aim of the study is to evaluate the effects of low-level laser therapy (LLLT) on patients with chronic periodontitis during a post-orthodontic period for 12 months. Following aspects will be assessed: 1. Effects on tooth stability maintenance and bone remodeling. 2. Effects on periodontal inflammation status. 3. Effects on cervical dentin sensitivity and quality of life. The study design is a randomised controlled trail. To eliminate any bias, the investigator will initially hypothesis there is no significant difference in the aforementioned aspects between teeth retained with an adjunctive LLLT strategy and those retained in a conventional regimen.

DETAILED DESCRIPTION:
The study design is a randomised split-mouth design based on the result of investigator's pilot study. Thirty-five non-smoking Ethnic Chinese patients (male and female, age: 25-65 years) with chronic periodontitis will be recruited. The teeth in experimental group will receive LLLT during orthodontic retention period for 12 months, while the teeth in the control (placebo) group will not receive laser therapy. Orthodontic occlusal indices will be measured to explore LLLT's role in maintaining tooth stability. The effects of LLLT on periodontal inflammation status will be evaluated by assessing clinical periodontal parameters and the levels of supra-gingival and sub-gingival bacteria. The effects of LLLT on bone remodelling will be explored by testing the biochemical biomarkers in gingival crevicular fluid (GCF). Cone-beam computed tomography will also be used to provide clinical evidence of periodontal status and bone remodelling. Possible effects of LLLT on patient's quality of life will be investigated via validated questionnaires, subjective assessment of tooth sensitivity, and objective measurement of bite force.

ELIGIBILITY:
Inclusion Criteria:

Thirty-five non-smoking Ethnic Chinese patients (male or female; age: 25-65 years) will be recruited from the Prince Philip Dental Hospital, Faculty of Dentistry, the University of Hong Kong into the following selection criteria:

1. Systemically health (with special regard to disease affecting tissue repair);
2. No medications required for periodontal therapy and no use of any antibiotic and/or anti-inflammatory medication in the preceding month;
3. Chronic periodontitis with at least two pairs (clinically matched) displaced single-rooted teeth (each pair of teeth is in the same arch but in two contralateral hemi-arches respectively belonging to the same tooth typology) having at least one site probing depth of 5 mm or more, interproximal attachment loss of 3 mm or more, and radiographic signs of alveolar bone loss before periodontal and orthodontic treatment.
4. Recent completion of orthodontic treatment and readiness for debonding and retainer delivery.

Exclusion Criteria:

1. smoking;
2. pregnancy;
3. under orthodontic treatment.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in probing pocket depth (PPD) | debond, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Record the changes of probing pocket depth in millimeters from baseline to 3 months, 6 months and 12 months through probing.
Changes in bleeding on probing (BOP) | debond, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Record the bleeding on probing changes from baseline to 3 months, 6 months and 12 months through probing.
Changes in clinical attachment loss (CAL) | debond, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Record the clinical attachment loss (CAL) changes from baseline to to 3 months, 6 months and 12 months.
Changes in plaque index (PI) | debond, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Record the plaque index (PI) changes from baseline to to 3 months, 6 months and 12 months.

SECONDARY OUTCOMES:
Orthodontic outcome stability | debond, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Assess the changes in Little's irregularity index (LII) in maxillar and mandibular anterior teeth in millimeters by measuring both plaster models and e-models
Alveolar bone remodelling | debond, 12 month follow-up
  Alveolar bone remodelling will be assessed by the changes in height (measured in millimeters) and thickness (measured in millimeters) of alveolar marginal bone surrounding predetermined target teeth according to Cone Beam computed tomography.
Supragingival and subgingival plaque | debond, 1 month follow-up, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Bacteria loads in supragingival and subgingival plaques will be recorded.
Cervical dentin sensitivity | debond, each week interval during the first months, 3 months, 6 months and 12 months
  Cervical dentin hypersensitivity will be evaluated by subjective assessment on a visual analogue scale (range from 0 to 100 mm) after a standardized stimuli applied on the test and control teeth.
Maximum voluntary bite force | debond, 1 month follow-up, 3 month follow-up, 6 month follow-up and 12 month follow-up
  Use an standardized occlusal force gauge to record the magnitude of bite force in newton (N).

CONTACTS AND LOCATIONS:
Overall Officials: Yanqi Yang, Principal Investigator — The Prince Philip Dental Hospital
Locations (1):
- The Prince Philip Dental Hospital, Hong Kong, Hong Kong